CLINICAL TRIAL: NCT03846297
Title: Optimisation of Decision Making for Defibrillator Implantation in Hypertrophic Cardiomyopathy
Acronym: OPTIM-HCM
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOR17412
Record Dates: First submitted 2019-02-04; First posted 2019-02-19 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: hypertrophic cardiomyopathy; implantable cardioverter defibrillator
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample of 30 ml will be collected at baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of the study is to improve implantable cardioverter defibrillator (ICD) implantation decision-making processing relevance by developing a new prediction model of sudden cardiac death (SCD) in hypertrophic cardiomyopathy (HCM), including newly identified potential biomarkers by magnetic resonance imaging (MRI) and genetics, through a prospective nationwide study, multivariate analysis and modelling of an absolute risk.

The secondary objective is to perform a medico-economic analysis of ICD implantation in order to define an optimal rule for ICD implantation in patients with HCM, taking into account the benefits of ICD, adverse effects of ICD and associated costs (cost of quality adjusted life years saved).

DETAILED DESCRIPTION:
HCM is a genetic disease, usually autosomal dominant, with a prevalence of about 1/500 in the general population. HCM represents a major cause of SCD in the young, and is the first cause of SCD in athletes less than 35 years of age. The only efficient prevention of SCD, apart from exercise restriction, is ICD.

Given this dreadful potential outcome of HCM, the identification of patients that should receive an ICD is of paramount importance. However, the indications for ICD are controversial and very different guidelines are currently available, coming from the American society of Cardiology, the French Haute Autorité de Santé and from the European society of Cardiology. In addition, these guidelines are all based on retrospective studies and have major limitations. The situation faces a critical need of improvement. Thus, this study has been designed with the objective to propose a revision of international recommendations for defibrillator implantation in HCM patients.

This prospective multicenter non-interventional single-arm study is planned to be conducted in 40 sites with a collection of clinical and biological data, carried out as required for the usual management and care of patients. No investigation will be performed specifically for this study except for an additional blood sample collection at baseline during routine outpatient care and annual interview during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of HCM based on conventional criteria (left ventricle wall thickness ≥ 15 mm in adult index or ≥ 13 mm in adult relatives) in the absence of abnormal loading conditions
* Aged ≥ 16 years
* Patient without or with a defibrillator (in this latter case it should have been implanted for primary prevention, not for secondary prevention)
* Affiliation to a social security insurance

Exclusion Criteria:

* Specific etiologies such as amyloidosis
* Patients with ICD as secondary prevention (after aborted SCD or sustained ventricular arrhythmia)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Inclusion of adults with HCM, as well as teenagers 16 or older since SCD occurs frequently in this age group
  * Necessary not to include specific etiologies such as amyloidosis because of a known different prognosis and natural history
  * Necessary not to include patients with ICD as secondary prevention because of a different prognosis and a worldwide consensus on the need for ICD implantation in this case
  * Necessary to include all cases whatever their date of diagnosis as the predictive modelling (primary objective) targets the actual population being followed up in real life, and will ultimately be applied on this population
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-09-23 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Improvement of the ability to predict major clinical events: C-index comparisons | throughout of the study, an average of 1 year
  Comparisons of the C-index obtained between with the new score and with the different existing scores or algorithms of actual processing used for ICD decision-making.
  C-index is a discrimination index, which will be determined after multivariate analyses and score modeling, in the case of the new score.
  This evaluate of the improvement of the ability to predict major clinical events during follow-up will toward to development of a new prediction model in patients with HCM in responding the main objective of the study.
  Data will be collected are: (composite end point): SCD, aborted sudden death, appropriate therapy of ICD that is a physiological equivalent of SCD.

SECONDARY OUTCOMES:
Cost-effectiveness study | throughout of the study, an average of 1 year
  To determine incremental cost-effectiveness ratio (ICER) of ICD decision, in order to assess the economic impact of defibrillator implantation as a function of the chosen rule for device implantation.
  Data will be collected are: direct costs (health insurance tariffs) of defibrillators, cost of their maintenance and for management of side effects, for the treatment of sudden death recovered, the medical transport, hospitalizations and for cardiology acts.
Cost-utility analysis | throughout of the study, an average of 1 year
  To determine incremental cost-utility ratio of ICD decision, in order to assess the economic impact of defibrillator implantation as a function of the chosen rule for device implantation.
  Data will be collected are: direct costs (health insurance tariffs) of defibrillators, cost of their maintenance and for management of side effects, for the treatment of sudden death recovered, the medical transport, hospitalizations and for cardiology acts.
Quality Adjusted Life Years | at baseline and at 6-year follow-up
  QALYs calculated using EQ-5d Index:
  "EQ5D-5L QoL questionnaire", a questionnaire established by EuroQol Group in 5 dimensions with 5 levers.
Improvement of the ability to predict major clinical events: C-index comparisons | at baseline
  Comparison of the C-index obtained between the new score developed for the primary objective and the C-index obtained when the following additional covariates are added to the multivariate predictive model: gender, maximum left ventricle wall thickness obtained by MRI, left atrial volume on echocardiography, left ventricle strain on echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CHARRON, MD, PhD, Principal Investigator — Centre de référence maladies cardiaques héréditaires, Hôpital Ambroise Paré & Hôpital Pitié-Salpêtrière
Locations (1):
- Centre de référence pour les cardiomyopathies et les troubles du rythme héréditaires ou rares - UF de Génétique, Hôpital Ambroise Paré,, Boulogne-Billancourt, Hauts-de-Seine, France

IPD SHARING:
Plan to Share IPD: No